CLINICAL TRIAL: NCT03864822
Title: Enhancing Inhibition With tDCS in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Danish National Research Foundation (Other)
Responsible Party: Principal Investigator, Megan McPhee, Principal Investigator, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: VN-20170034-v5
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Stimulation type will be randomized by a colleague not involved in the study. A single investigator will assess all outcomes on all participants before and after each phase of stimulation, but participants not the investigator will be aware of Active/Sham assignment until after study completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): 30s ramp to 2mA with 20 minute session of active High-Definition Transcranial Direct Current Stimulation at 2mA
  Interventions: Device: High-Definition Transcranial Direct Current Stimulation
- Sham tDCS (Placebo Comparator): 30s ramp to 2mA with High-Definition Transcranial Direct Current Stimulation, then device stops stimulating for 20 minutes
  Interventions: Device: High-Definition Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High-Definition Transcranial Direct Current Stimulation — Device uses an array of electrodes over the scalp, in contact via gel, to provide a weak electrical current.

SUMMARY:
This cross-over study intends to use consecutive days of active versus sham transcranial direct current stimulation (tDCS) to enhance descending inhibition and look at resulting clinical effects in people with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy men and women
* Aged 18-60 years
* Continuous pain (>3days pain/week) episode lasting at least 3 months, sufficient to limit daily activities
* Pain in the region posteriorly between the inferior border of the 12th rib and the lower gluteal fold (low back pain) at the time of recruitment
* Able to speak, read and understand English

Exclusion Criteria:

* Pregnancy
* Low back pain associated with menstruation
* Currently seeking active treatment for low back pain
* Red flags symptoms (i.e. fever, malaise, progressive neurologic deficit, significant trauma, prolonged corticosteroid use or osteoporosis, pain worst at night, urinary or faecal incontinence, or unintended weight loss)
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Current or previous neurologic, musculoskeletal, mental, or other illnesses which may affect the trial
* Current or previous chronic or recurrent pain condition other than low back pain
* Current regular use of analgesic medication or other medication which may affect the trial
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | Day 0 (Pre) to Day 3 (Post) in each stimulation phase
  Change in cuff pain threshold with contralateral cuff conditioning stimulus

SECONDARY OUTCOMES:
Temporal Summation of Pain | Day 1 (Pre) to Day 3 (Post) in each stimulation phase
  Change in pain intensity ratings (i.e. on an electronic Visual Analogue Scale from 0=no pain to 10=worst pain imaginable) across series of 10 x 1s cuff stimuli at 0.5Hz (scores are normalized to first rating by subtraction and grouped into 3 epochs of 3 inflations with higher change scores indicating higher summation/facilitation)
Pressure Pain Thresholds | Day 1 (Pre) to Day 3 (Post) in each stimulation phase
  Handheld algometry over the extensor carpi radialis, upper trapezius, lower back and gastrocnemius muscles
Pain Intensity | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  Visual Analogue Scale from 0=no pain to 10=worst pain imaginable currently at rest and with worst movement, as well as maximum in past week
Pain Unpleasantness | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  Visual Analogue Scale from 0=not unpleasant at all to 10=most unpleasant sensation imaginable currently at rest and with worst movement, as well as maximum in past week
Pain Area | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  Total number of pixels coloured on an electronic body chart (Navigate Pain)
Roland-Morris Disability Questionnaire | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  Measures back-related disability for 24 statements of potentially afflicted tasks with dichotomous responses. Minimum 0 to maximum 24 with higher scores indicating worse disability.
Back Performance Scale | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  5 Task scale rated as per performance as a functional measure of back-related disability (each task is rated on a 4 point Likert scale 0-3 and summed to give total), scored from 0-15 with higher scores indicating more pain and dysfunction during task performance. Here will be used to characterize functional disability.

OTHER OUTCOMES:
Flanker Task Learning | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  Reaction time to selective attention based computer task
Affect Manipulation | Day 0 (Pre) to Day 3 (Post) and 2 weeks post for each stimulation phase
  Effect of image watching on ratings of mood and arousal. Mood and arousal will be measured with the Self Assessment Manikin - a 9 point Likert-type scale with 1 representing most negative/most calm, 5 as neutral, and 9 as most positive/most aroused.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E McPhee, BPhty MSc, Principal Investigator — Center for Neuroplasticity and Pain (CNAP), SMI, Aalborg University
Locations (1):
- CNAP, SMI, Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after study completion and publication in necessary cases on request

REFERENCES:
- [Derived] McPhee ME, Graven-Nielsen T. Medial Prefrontal High-Definition Transcranial Direct Current Stimulation to Improve Pain Modulation in Chronic Low Back Pain: A Pilot Randomized Double-blinded Placebo-Controlled Crossover Trial. J Pain. 2021 Aug;22(8):952-967. doi: 10.1016/j.jpain.2021.02.012. Epub 2021 Mar 4. PMID 33676009